CLINICAL TRIAL: NCT01079468
Title: Cognition in Postoperative Total Hip Arthroplasty and Total Hip Resurfacing Patients
Status: Completed | Type: Observational
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: William Hozack, MD, Prinicple Investigator, Rothman Institute
Other Study IDs: RIUHOZ 10-01
Record Dates: First submitted 2010-03-01; First posted 2010-03-03 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Cognition
Keywords: Transient cognitive decline following orthopaedic surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Total Hip Arthroplasty
- Total Hip Resurfacing Arthroplasty

SUMMARY:
Transient cognitive changes after surgery may be due to many different factors. It is estimated that between 5-29% of patients undergoing orthopedic surgery experience a transient decline in their cognition. Fat and bone marrow debris embolization can cause cognitive changes if they enter the cerebral circulation in significant numbers. During total hip arthroplasty the placement of the femoral stem leads to a rise in intramedullary pressure which can cause fat and bone marrow debris to embolize into the systemic circulation. Total hip resurfacing arthroplasty avoids entrance into the femoral canal. The purpose of this study is to assess transient cognitive changes after total hip arthroplasty and compare them to patients undergoing total hip resurfacing arthroplasty. We hypothesize that patients undergoing total hip resurfacing arthroplasty will experience less transient cognitive changes due to the avoidance of violating the femoral canal during the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Male and non-pregnant, non-lactating, female subjects who are 18 and older
2. Subjects who are able and willing to provide informed consent
3. Subjects deemed able to comply with study schedule visits and procedures
4. Subjects undergoing elective THA procedures
5. Subjects undergoing elective total hip resurfacing arthroplasty
6. Subjects in satisfactory health as determined by the investigator on the basis of medical history and physical examination.

Exclusion Criteria:

1. Subjects with or with a history of Parkinson's Disease
2. Subjects with a history of depression as reported in their past medical history
3. Subjects with a history of dementia as reported in their past medical history
4. Subjects currently using antidepressants
5. Subjects currently using antipsychotic medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing either Total Hip Arthroplasty or Total Hip Resurfacing Arhtroplasty at our Institution
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Degree of transient cognitive changes postoperatively as measured by the Folstein mini-mental examination

SECONDARY OUTCOMES:
Percentage of patient who experience transient cognitive decline following Total Hip Arthroplasty or total hip resurfacing arthroplasty as measured by the Folstein mini-mental examination

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Koch S, Forteza A, Lavernia C, Romano JG, Campo-Bustillo I, Campo N, Gold S. Cerebral fat microembolism and cognitive decline after hip and knee replacement. Stroke. 2007 Mar;38(3):1079-81. doi: 10.1161/01.STR.0000258104.01627.50. Epub 2007 Jan 25. PMID 17255544
- [Background] Koessler MJ, Pitto RP. Fat embolism and cerebral function in total hip arthroplasty. Int Orthop. 2002;26(5):259-62. doi: 10.1007/s00264-002-0380-2. Epub 2002 Jun 25. No abstract available. PMID 12378348